CLINICAL TRIAL: NCT07318207
Title: A Pragmatic Clinical Trial of Time-restricted Eating in the University of Kentucky Barnstable Brown Diabetes Center
Brief Title: Time-restricted Eating for Patients With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Justin (Matt) Thomas (Other)
Responsible Party: Sponsor-Investigator, Justin (Matt) Thomas, Postdoctoral Fellow, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105493; Funding Organization (Other: University of Kentucky Barnstable Brown Diabetes and Obesity Center)
Record Dates: First submitted 2025-12-22; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-restricted eating (Experimental): Subjects in this group will consume all daily calories within a 10-h window during the day for 1-year.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Subjects will consume all daily calories within a 10-hour (10h +/- 1hr) window during the daytime, ending by 8:00pm. Subjects will text the time of their first and last daily calorie intake for the duration of the study.

SUMMARY:
This is a single-arm pragmatic clinical trial of time-restricted eating in patients with type 2 diabetes. Patients will be recruited from the University of Kentucky Barnstable Brown Diabetes Center. Subjects will participate in a 10-hour time-restricted eating intervention for 1-year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes

Exclusion Criteria:

* Pregnant or breastfeeding
* Diagnosed eating disorder
* Night shift worker
* Taking drugs which induce hypoglycemia
* Unable or unwilling to participate in the time-restricted eating intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | At least 2 timepoints between baseline and 1 year. Since labs will depend on clinic visits, exact timeframe will vary.
  HbA1c data will be gathered from patient charts from routine labs collected during clinic visits.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index | Baseline, 6 months, and 1 year
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index and will be reported as a composite score ranging from 0 to 21 with a higher score indicating worse sleep quality.
Change in Short Form-36 Quality of Life questionnaire scores | Baseline, 6 months, and 1 year
  Quality of life will be collected using the Short Form-36 Quality of Life questionnaire and scores for 8 scales will be analyzed: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores for each scale will range from 0 to 100 with higher scores indicating more favorable health.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Thomas, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Barnstable Brown Diabetes Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No